CLINICAL TRIAL: NCT05826704
Title: Exploring the Effects of Lactobacillus Paracasei PS23 on Workplace-related Stress Symptoms Among Office Workers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The company had to re-decorate
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 22CT044be
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Stress
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PS23 (Experimental): 2 capsule daily
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): 2 capsule daily
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Participants will be taking 2 capsule a day for 6 weeks

SUMMARY:
A total of 120 subjects are expected to be recruited over a 3-year period starting after IRB approval, divided into two groups of 60 subjects, receiving PS23 or placebo, and completing a 6-week trial period.

DETAILED DESCRIPTION:
There is still a lack of research to explore the interaction between high-pressure workers and probiotics to improve the intestinal microbiota and further affect its relationship with sleep, inflammation, and anti-oxidation, and further studies are still needed to confirm the clinical effect. A total of 120 subjects are expected to be recruited over a 3-year period starting after IRB approval, divided into two groups of 60 subjects, receiving PS23 or placebo, and completing a 6-week trial period.

ELIGIBILITY:
Inclusion Criteria:

1. Administrative staff of JARLLYTEC CO., LTD.
2. Age 20-65 years old
3. Those who feel that they are in a medium to high stress situation

Exclusion Criteria:

1. Have taken antibiotics within one month or are receiving antibiotic treatment
2. Have taken probiotic products within two weeks (excluding yogurt, yogurt, Yakult and other related foods)
3. have a history of cancer
4. Those who are allergic to lactic acid bacteria products
5. Those who are currently taking medication for acute illness, mental illness or sleep disorder
6. Pregnant or breastfeeding
7. The project host judges that it is not suitable to participate in the researcher

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale, PSS | From Baseline to 6 Weeks Assessed
  The PSS scores is a rating tool used to gauge the course of stress. The minimum total score possible is 0 and the maximum total score possible is 56. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Insomnia Severity Index, ISI | From Baseline to 6 Weeks Assessed
  The ISI is a rating tool used to gauge of sleeping. Higher values represent a worse outcome. The minimum total score possible is 0 and the maximum total score possible is 28. Higher values represent a worse outcome.
The State-Trait Anxiety Inventory, STAI | From Baseline to 6 Weeks Assessed
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). The minimum total score possible is 40 and the maximum total score possible is 160. Higher scores indicate greater anxiety.
Patient Health Questionnaire, PHQ-9 | From Baseline to 6 Weeks Assessed
  Measure for Major Depressive Disorder from questionnaire responses, clinically significant depression defined as a PHQ-9 score of equal to or greater than 10.
The Quality of Life, Enjoyment, and Satisfaction Questionnaire-Short Form-16, QLESQ-16 | From Baseline to 6 Weeks Assessed
  The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16 (QLESQ-16) is a valid, reliable self-report instrument for assessing quality of life. The minimum total score possible is 14 and the maximum total score possible is 70. The higher score the better satisfaction.
VAS-GI | From Baseline to 6 Weeks Assessed
  Visual Analogue Scale for GI symptoms, VAS-GI (visual analogue scale, VAS 0-10) was designed to measure the response of symptoms and well-being in patients after taking probiotics.
Brief Fatigue Inventory | From Baseline to 6 Weeks Assessed
  Brief Fatigue Inventory（ BFI）is a nine item scale used to evaluate the intensity of fatigue and the interference of fatigue to normal activities. The classification of fatigue severity is: Mild fatigue (1-3), Moderate fatigue (4-6) and Severe fatigue (7-10).
Patient Global Impression scales of Improvement rated by patient, PGI-C | From Baseline to 6 Weeks Assessed
  The PGIC is a single-item questionnaire that asks the patient to assess their TD symptoms at specific visits after initiating therapy. The PGIC uses a 7 point Likert Scale, ranging from very much worse (-3) to very much improved (+3), to assess overall response to therapy.
Saliva Cortisol | From Baseline to 6 Weeks Assessed
  Cortisol is a steroid hormone that is produced by the adrenal glands which sit on top of each kidney. When released into the bloodstream, cortisol can act on many different parts of the body and can help:
  body respond to stress or danger increase your body's metabolism of glucose control your blood pressure reduce inflammation. Cortisol is also needed for the fight or flight response which is a healthy, natural response to perceived threats. The amount of cortisol produced is highly regulated by your body to ensure the balance is correct.
Saliva α-amylase | From Baseline to 6 Weeks Assessed
  Salivary alpha-amylase activity (sAA) is often considered to be surrogate markers of sympathetic activation in response to stress.
Saliva IgA | From Baseline to 6 Weeks Assessed
  Secretory IgA in saliva stands in a negative correlation to the level of the experienced stress
Saliva Lactoferrin | From Baseline to 6 Weeks Assessed
  lactoferrin's multiple activities lie in its capacity to bind iron and to interact with the molecular and cellular components of hosts and pathogens. it can bind and sequester lipopolysaccharides, thus preventing pro-inflammatory pathway activation, sepsis and tissue damages.
Saliva Lysozyme | From Baseline to 6 Weeks Assessed
  Lysozyme plays a pivotal role in the prevention of bacterial infections by attacking peptidoglycan in the bacterial cell wall.
Job Stress Scale from the Ministry of Labor | From Baseline to 6 Weeks Assessed
  The job stress scale from Ministry of Labor is a rating tool used to gauge of stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wu SI, Kao KL, Lin CJ, Lin YJ, Lin IC, Chen WL. Effect of lacticaseibacillus paracasei PS23 on anxiety and sleep difficulties among office workers: a double-blind, randomized controlled pilot trial. Ann Gen Psychiatry. 2025 Oct 9;24(1):59. doi: 10.1186/s12991-025-00599-1. PMID 41068940